CLINICAL TRIAL: NCT07146568
Title: Evaluating the Implementation and Effectiveness of the Pink and Pearl Campaign on Lung Cancer Screening at Christian Hospital
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 202508075
Record Dates: First submitted 2025-08-21; First posted 2025-08-28 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Lung Cancer; Cancer of the Lung
Keywords: Lung cancer screening (LCS); Pink and Pearl Campaign; Breast cancer screening (BCS); Low-dose computed tomography (LDCT); Smoking history; Health disparities; Screening behavior; Feasibility; Acceptability; Appropriateness
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Participants - scheduled for mammography and eligible for LCS (Experimental): All women coming in for breast cancer screening will be assessed for LCS eligibility using a screening questionnaire administered by mammography technicians. Patients who are determined to be eligible for LCS will be asked by the mammography technician if they will opt into being contacted by the nurse navigator, who will facilitate their referral to primary care to schedule a LCS appointment at Siteman Cancer Center.
  Interventions: Other: Pink and Pearl Campaign
- Providers (No Intervention): Providers in the breast radiology service who referred women to LCS. Investigators will gather information on the feasibility, acceptability, and appropriateness of the Pink and Pearl project.

INTERVENTIONS:
Other: Pink and Pearl Campaign — This campaign leverages established infrastructure such as nurse navigation and referral to screening or primary care for further shared decision-making on cancer screening.
  Arms: Participants - scheduled for mammography and eligible for LCS

SUMMARY:
Inspired by the ongoing Pink & Pearl Campaign, the breast radiology service of Christian Hospital in north St. Louis County will partner with Siteman Cancer Center to pilot this campaign in its mammography clinics in order to promote awareness, referral, and completion of lung cancer screening (LCS) among eligible women. This campaign leverages established infrastructure such as nurse navigation and referral to screening or primary care for further shared decision-making on cancer screening. The purpose of this study is to evaluate the effectiveness of the Pink & Pearl Campaign in improving LCS uptake among LCS-eligible women undergoing mammography at Christian Hospital. This evaluation is grounded in the Integrated Screening Action Model that depicts individual- and environmental-level influences on the screening behavior process. Using an explanatory sequential mixed methods design, which combines both quantitative and qualitative approaches, our specific aims for this proposal are to: a) assess whether the Pink & Pearl Campaign increases referrals and uptake/completion of LCS among LCS-eligible women undergoing screening mammography; b) determine median time-to-screening after referral to LCS; and c) evaluate individual and health system factors influencing LCS uptake and implementation outcomes of the campaign. These implementation outcomes will help identify whether the campaign was put in place successfully or not. This proposal will inform strategies for integrating cancer screening programs to improve poorly performing programs like LCS.

ELIGIBILITY:
Eligibility Criteria - Interventional Study

* Undergoing screening mammography at Christian Hospital
* Between the ages of 50-80 years (inclusive)

Eligibility Criteria - Survey and Interview Sub-Studies

* Part of the interventional study
* Reporting a 20 pack-year equivalent of either current smoking history or have quit in the past 15 years
* Can speak and understand English
* Not diagnosed with a serious health problem that will limit life expectancy (such as previous history of lung cancer, symptoms of lung cancer such as hemoptysis or unexplained weight loss of more than 6.8 kg (15 lb) in the previous year)
* Willing and able to get treatment if lung cancer is found
* Able to understand and willing to sign an IRB-approved written informed consent document

Eligibility Criteria - Providers

* At least 20 years of age
* Involved in the breast radiology service or referred at least one patient to the Pink & Pearl Campaign
* Able to provide verbal consent to participate in the interview

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 5515 (Estimated)
Dates: Start 2026-02-16 (Estimated); Primary Completion 2026-08-31 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of women referred from the breast radiology service who successfully complete LCS 6-months post-Pink & Pearl implementation | At 6 months
  The investigators will compare the baseline prevalence of LCS among women undergoing BCS to the prevalence of LCS among women undergoing BCS 6 months after implementation of the Pink & Pearl Campaign.

SECONDARY OUTCOMES:
Median time-to-screening | At 6 months
  The investigators will compare differences in time-to-lung cancer screening across heterogenous populations
Acceptability of Pink & Pearl Campaign | At 6 months
  Defined as the perception that the campaign is agreeable or satisfactory

OTHER OUTCOMES:
Number of individual level barriers to LCS completion | At 6 months
Number of health system level barriers to LCS completion | At 6 months
Feasibility of Pink & Pearl Campaign | At 6 months
  Defined as extent to which strategy is suitable for a routine use in a setting
Appropriateness of Pink & Pearl Campaign | At 6 months
  Defined as perceived fit, relevance or compatibility of the strategy or practice for a given setting

CONTACTS AND LOCATIONS:
Overall Officials: Beryne Odeny, M.D., MPH, Ph.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Barnes-Jewish Christian Hospital, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: Yes
Plan to share results interpretations.
Supporting Information: Study Protocol, SAP
Time Frame: For a period of 1 year.
Access Criteria: Contact the Principal Investigator or Central Contact Back-up via email.

REFERENCES:
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu